CLINICAL TRIAL: NCT02113839
Title: Breathlessness Perception in COPD: Relationship With Exacerbation Frequency
Brief Title: Dyspnea in COPD: Relationship With Exacerbations Frequency
Acronym: DPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Isabel Blanco, MD, PhD, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DysPerEx
Record Dates: First submitted 2014-04-04; First posted 2014-04-15 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2014-04

CONDITIONS: Dyspnea
Keywords: Dyspnea perception; COPD; Exacerbations; CO2 rebreathing test
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive | interventions — Ventilation; Inspiratory Capacity; Carboxyhemoglobin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No frequent exacerbators (Active Comparator): Patients without exacerbations: 0 or 1 that did not required hospitalization in the previous year.
  Interventions:
  * Spirometry
  * Emogas analysis
  * Modified Borg Dyspnea Scale
  * CO Exhaled breath
  * P01
  * FeNO
  Interventions: Procedure: Spirometry; Procedure: CO Exhaled breath; Procedure: P01; Procedure: FeNO
- Frequent exacerbators (Active Comparator): Patients with frequent exacerbations: ≥2 or ≥1 if it required hospitalization in the previous year.
  Interventions:
  * Spirometry
  * Emogas analysis
  * Modified Borg Dyspnea Scale
  * CO Exhaled breath
  * P01
  * FeNO
  Interventions: Procedure: Spirometry; Procedure: CO Exhaled breath; Procedure: P01; Procedure: FeNO

INTERVENTIONS:
Procedure: Spirometry — Before re-breathing (if the patient not performed one 6 months in advance).
  Other Names: FEV1; FVC; FEV1/FVC; VC; TLC; Rwc; DLCO; DLCO/VA; Ventilation (VE); Inspiratory capacity (IC)
Procedure: CO Exhaled breath — In current smokers of both arms to confirm that the patient has not smoked in the past three hours and to asses the smoking status (heavy, moderate, light).
  Other Names: CO (ppm); COHb (%)
Procedure: P01 — P01 is the negative airway pressure generated during the ﬁrst 100 ms of an occluded inspiration. It's an estimation of the neuromuscular drive to breathe.
Procedure: FeNO — The measurement of fraction of exhaled nitric oxide during exacerbations of COPD is higher than normal.

SUMMARY:
The perception of breathlessness varies significantly among COPD patients with similar severity of airflow limitation; those with poorer perception report less exacerbations as compared to those with frequent exacerbations.

Cross-sectional comparison of breathlessness perception in COPD patients with frequent exacerbations or without frequent exacerbations.

To assess "Breathlessness Perception" the investigators will increase the ventilatory demand of the patients by CO2-rebreathing method.

DETAILED DESCRIPTION:
The perception of breathlessness varies between individuals. This is a well-established concept in asthma, but mostly unexplored in COPD; the relationship between airflow limitation (FEV1, % ref.) and breathlessness (mMRC) is weak.

The perception of breathlessness varies significantly among COPD patients with similar severity of airflow limitation; those with poorer perception report less exacerbations as compared to those with frequent exacerbations.

It is a cross-sectional comparison of breathlessness perception in COPD patients with frequent exacerbations (≥2 or ≥1 with hospitalization in the previous year) or without frequent exacerbations (0 or 1 without hospitalization in the previous year).

To assess "Breathlessness Perception" the investigators will increase the ventilatory demand of the patients by CO2-rebreathing method. CO2 rebreathing test will be conducted to evaluate the acute ventilatory response to CO2 inhalation used to estimate central chemoreceptor responsiveness in patients with the obstructive pulmonary disease.

Simple descriptive statistics (unpaired T-test) and correlation analysis (bivariate and multivariate) will be used to analyze results.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of COPD (Gold 2 or 3 or 4)
* >2 months from last exacerbation and no change in therapy

Exclusion Criteria:

* patients on regular sedative drugs
* patients with neuromuscular diseases
* patients with respiratory failure and/or in long-term oxygen therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The negative airway pressure generated during the ﬁrst 100 ms of an occluded inspiration, which is an estimation of the neuromuscular drive to breathe. (P01 ) | Baseline

SECONDARY OUTCOMES:
Borg scale | Baseline
  10-point subjective scoring system, in which a patient rates his/her effort of exertion.
Fractional exhaled nitric oxide (FeNO) | Baseline
Inspiratory capacity (IC) | Baseline
  The sum of inspiratory reserve volume and tidal volume.
Ventilation at rest | Baseline
CO exhaled test | Baseline
  Testing for Carbon Monoxide in exhaled breath in current smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Blanco Vich, MD, PhD, Principal Investigator — Hospital Clínic; Alvar G Agustí, MD, PhD, Study Director — Hospital Clínic
Locations (1):
- Hospital Clínic, Barcelona, BCN, Spain

REFERENCES:
- [Background] Davis SQ, Permutt Z, Permutt S, Naureckas ET, Bilderback AL, Rand CS, Stein BD, Krishnan JA. Perception of airflow obstruction in patients hospitalized for acute asthma. Ann Allergy Asthma Immunol. 2009 Jun;102(6):455-61. doi: 10.1016/S1081-1206(10)60117-2. PMID 19558002
- [Background] Miravitlles M, Anzueto A, Legnani D, Forstmeier L, Fargel M. Patient's perception of exacerbations of COPD--the PERCEIVE study. Respir Med. 2007 Mar;101(3):453-60. doi: 10.1016/j.rmed.2006.07.010. Epub 2006 Aug 30. PMID 16938447
- [Background] Agusti A, Calverley PM, Celli B, Coxson HO, Edwards LD, Lomas DA, MacNee W, Miller BE, Rennard S, Silverman EK, Tal-Singer R, Wouters E, Yates JC, Vestbo J; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) investigators. Characterisation of COPD heterogeneity in the ECLIPSE cohort. Respir Res. 2010 Sep 10;11(1):122. doi: 10.1186/1465-9921-11-122. PMID 20831787
- [Background] Garcia-Aymerich J, Gomez FP, Benet M, Farrero E, Basagana X, Gayete A, Pare C, Freixa X, Ferrer J, Ferrer A, Roca J, Galdiz JB, Sauleda J, Monso E, Gea J, Barbera JA, Agusti A, Anto JM; PAC-COPD Study Group. Identification and prospective validation of clinically relevant chronic obstructive pulmonary disease (COPD) subtypes. Thorax. 2011 May;66(5):430-7. doi: 10.1136/thx.2010.154484. Epub 2010 Dec 21. PMID 21177668
- [Background] Fan VS, Gaziano JM, Lew R, Bourbeau J, Adams SG, Leatherman S, Thwin SS, Huang GD, Robbins R, Sriram PS, Sharafkhaneh A, Mador MJ, Sarosi G, Panos RJ, Rastogi P, Wagner TH, Mazzuca SA, Shannon C, Colling C, Liang MH, Stoller JK, Fiore L, Niewoehner DE. A comprehensive care management program to prevent chronic obstructive pulmonary disease hospitalizations: a randomized, controlled trial. Ann Intern Med. 2012 May 15;156(10):673-83. doi: 10.7326/0003-4819-156-10-201205150-00003. PMID 22586006
- [Background] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Background] Rodriguez-Roisin R. Toward a consensus definition for COPD exacerbations. Chest. 2000 May;117(5 Suppl 2):398S-401S. doi: 10.1378/chest.117.5_suppl_2.398s. PMID 10843984
- [Background] Seemungal TA, Donaldson GC, Bhowmik A, Jeffries DJ, Wedzicha JA. Time course and recovery of exacerbations in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2000 May;161(5):1608-13. doi: 10.1164/ajrccm.161.5.9908022. PMID 10806163
- [Background] Jones PW, Nadeau G, Small M, Adamek L. Characteristics of a COPD population categorised using the GOLD framework by health status and exacerbations. Respir Med. 2014 Jan;108(1):129-35. doi: 10.1016/j.rmed.2013.08.015. Epub 2013 Aug 30. PMID 24041746
- [Background] Agusti AG, Villaverde JM, Togores B, Bosch M. Serial measurements of exhaled nitric oxide during exacerbations of chronic obstructive pulmonary disease. Eur Respir J. 1999 Sep;14(3):523-8. doi: 10.1034/j.1399-3003.1999.14c08.x. PMID 10543270
- [Background] Parker J, Wolansky LJ, Khatry D, Geba GP, Molfino NA. Brain magnetic resonance imaging in adults with asthma. Contemp Clin Trials. 2011 Jan;32(1):86-9. doi: 10.1016/j.cct.2010.09.006. Epub 2010 Sep 18. PMID 20854931
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Derived] Scioscia G, Blanco I, Arismendi E, Burgos F, Gistau C, Foschino Barbaro MP, Celli B, O'Donnell DE, Agusti A. Different dyspnoea perception in COPD patients with frequent and infrequent exacerbations. Thorax. 2017 Feb;72(2):117-121. doi: 10.1136/thoraxjnl-2016-208332. Epub 2016 Sep 1. PMID 27586869